CLINICAL TRIAL: NCT02632656
Title: Plasma ExtrAcellular RNAs and Biomarkers of Heart FaiLure During Decongestion: PEARL-HF Study
Acronym: PEARL-HF
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Saumya Das, Physician, Massachusetts General Hospital
Other Study IDs: 2015P001658
Record Dates: First submitted 2015-12-11; First posted 2015-12-17 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood collected at various time points during CHF therapy, processed for ex-RNAs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with congestive heart failure: Patients with congestive heart failure (CHF) who are followed in the hospital or clinic setting, with optimization of medical therapy
  Interventions: Other: Monitoring on heart failure therapy

INTERVENTIONS:
Other: Monitoring on heart failure therapy — This is a prospective observational study where participants will have serial blood collection on medical therapy for heart failure.

SUMMARY:
The primary objective is to measure the association between extracellular RNA (ex-RNA) levels in plasma in patients receiving aggressive outpatient therapy for CHF with (1) cardiac remodeling and (2) cardiovascular events. The investigators will follow patients during standard medical therapy for CHF to assess changes in ex-RNA levels in the plasma, and how these are associated with cardiac remodeling (by cardiac imaging) and outcomes.

DETAILED DESCRIPTION:
Nearly 5 million people in the United States have congestive heart failure (CHF). Although medical therapy such as beta-blockers, angiotensin converting enzyme (ACE) inhibitors, angiotensin-receptor blockers (ARBs) and aldosterone antagonists has improved prognosis, the overall rate of hospital admissions has continued to rise in the last decade and the mortality for patients with symptomatic heart failure remains worse than the majority of cancers in this country. Accordingly, significant opportunities exist for the improvement in outcomes of patients with CHF, both from a morbidity and mortality standpoint. Such opportunities may lie in the outpatient medical management of patients with CHF.

In this study, the primary objective is to measure the association between extracellular RNA (ex-RNA) levels in plasma in patients receiving aggressive outpatient therapy for CHF with (1) cardiac remodeling and (2) cardiovascular events. The investigators will follow patients during standard medical therapy for CHF to assess changes in ex-RNA levels in the plasma, and how these are associated with cardiac remodeling (by cardiac imaging) and outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 21 years of age
2. Left ventricular ejection fraction ≤ 50% (at any time in the past)
3. Symptomatic (NYHA class II-IV) heart failure (as diagnosed by clinician, radiographic images, or abnormal natriuretic peptide level)
4. Hospital admission, Emergency Department visit, or outpatient diuretic escalation of therapy for destabilized HF at least once in the 6 months prior to enrollment

Exclusion Criteria:

1. Severe renal insufficiency defined as serum creatinine > 2.5 mg/dl
2. United Organ Network Sharing status 1B for heart transplantation (outpatient inotrope use, LV assist device)
3. Inoperable aortic valvular heart disease
4. Life expectancy <1 year due to causes other than HF such as advanced cancer
5. Cardiac transplantation or revascularization indicated or expected within 6 months
6. Severe obstructive or restrictive pulmonary disease, defined as a forced expiratory volume in 1 sec <1 L (when diagnosed as standard of care)
7. Subject unable or unwilling to provide written informed consent
8. Coronary revascularization (percutaneous coronary intervention or bypass surgery) within the previous 3 months

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 200 eligible subjects. These subjects will be enrolled from the Massachusetts General Heart Failure Center population, from the Yawkey Center for Outpatient Care, upon discharge from the inpatient services at Massachusetts General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-12; Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to death | 24 months
Time to decompensated heart failure (HF) requiring in-patient admission or ER visit or IV diuretic therapy in the outpatient realm | 24 months
  • New onset of classic symptoms and signs of destabilized HF, including lower extremity edema, jugular venous distension, bibasilar crackles, orthopnea and paroxysmal nocturnal dyspnea
Time to acute coronary syndrome | 24 months
  Myocardial infarction
Time to stroke or transient ischemic attack | 24 hours
Time to ventricular arrhythmia | 24 months
  Clinically significant ventricular arrhythmia, defined as ventricular arrhythmia plus one of the following:

SECONDARY OUTCOMES:
Change in left ventricular (LV) end-systolic volume (in %) | 12 months
Change in LV ejection fraction (%) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States